CLINICAL TRIAL: NCT05596149
Title: Assessment of the Cytotoxic and Genotoxic Effect of Toothpastes With Different Forms of Fluoride on the Buccal Mucosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zagreb (Other)
Collaborators: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Jasen Vladislavić, Pulmonology Resident, Medical Doctor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2181-198-03-04-22-0003
Record Dates: First submitted 2022-10-04; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: DNA Damage
Keywords: Fluoride; Toothpaste; Cytotoxicity; Genotoxicity; Buccal mucosa; DNA damage
MeSH Terms: interventions — Toothpastes; Fluorides; Sodium Fluoride; fluorophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Toothpaste without fluoride (Active Comparator): A group of participants that will be using toothpaste without fluoride.
  Interventions: Other: Toothpaste without fluoride
- Toothpaste with sodium fluoride (Experimental): A group of participants that will be using toothpaste with sodium fluoride.
  Interventions: Other: Toothpaste with sodium fluoride
- Toothpaste with sodium monofluorophosphate (Experimental): A group of participants that will be using toothpaste with sodium monofluorophosphate.
  Interventions: Other: Toothpaste with sodium monofluorophosphate
- Toothpaste with amine fluoride (Experimental): A group of participants that will be using toothpaste with amine fluoride.
  Interventions: Other: Toothpaste with amine fluoride

INTERVENTIONS:
Other: Toothpaste without fluoride — A sample of cells from the area of the buccal mucosa of each of the subjects will be taken with a cytological brush just before the start of using the toothpaste without fluoride and 30, 45 and 60 days after the start of use. Cell suspension is applied on a microscopy slide. Slides will be stained with Fast Green FCF dye and analyzed with an epifluorescence microscope. After using each tested toothpaste, the respondents will be given a specially designed questionnaire with questions related to their opinion about the used oral hygiene product.
  Arms: Toothpaste without fluoride
Other: Toothpaste with sodium fluoride — A sample of cells from the area of the buccal mucosa of each of the subjects will be taken with a cytological brush just before the start of using the toothpaste with sodium fluoride and 30, 45 and 60 days after the start of use. Cell suspension is applied on a microscopy slide. Slides will be stained with Fast Green FCF dye and analyzed with an epifluorescence microscope. After using each tested toothpaste, the respondents will be given a specially designed questionnaire with questions related to their opinion about the used oral hygiene product.
  Arms: Toothpaste with sodium fluoride
Other: Toothpaste with sodium monofluorophosphate — A sample of cells from the area of the buccal mucosa of each of the subjects will be taken with a cytological brush just before the start of using the toothpaste with sodium monofluorophosphate and 30, 45 and 60 days after the start of use. Cell suspension is applied on a microscopy slide. Slides will be stained with Fast Green FCF dye and analyzed with an epifluorescence microscope. After using each tested toothpaste, the respondents will be given a specially designed questionnaire with questions related to their opinion about the used oral hygiene product.
  Arms: Toothpaste with sodium monofluorophosphate
Other: Toothpaste with amine fluoride — A sample of cells from the area of the buccal mucosa of each of the subjects will be taken with a cytological brush just before the start of using the toothpaste with amine fluoride and 30, 45 and 60 days after the start of use. Cell suspension is applied on a microscopy slide. Slides will be stained with Fast Green FCF dye and analyzed with an epifluorescence microscope. After using each tested toothpaste, the respondents will be given a specially designed questionnaire with questions related to their opinion about the used oral hygiene product.
  Arms: Toothpaste with amine fluoride

SUMMARY:
The remarkable therapeutic anticaries effect of fluoride is well recognized, but in recent years, toxic effects on the oral mucosa have been discussed. So far, many in vivo studies examining the genotoxic and cytotoxic effect of fluoride in human cells (lymphocytes, bone marrow, germ cells) have been carried out, but there are no studies examining the effect of fluoride on cells of the buccal mucosa. In vitro studies have shown that sodium fluoride can be toxic to fibroblasts of the oral mucosa by inhibiting protein synthesis, suppressing mitochondrial function and consequently reducing the amount of intracellular ATP.

The study would include 80 participants, aged between 18 and 75. All subjects would use the same toothpaste without fluoride for the first month, and then they would be randomly divided into four groups, where three groups would receive a toothpaste with fluoride with one of the active substances (sodium fluoride, sodium monofluorophosphate, amine fluoride) for the next 60 days, while the control group would continue to use the toothpaste without fluorine. Swabs of the buccal mucosa would be taken at 0 (before the start of use) and 30, 45 and 60 days after the start of using the tested toothpastes.

The aim of this research would be to examine the cytotoxic and genotoxic effect of toothpastes containing fluoride with different active substances and to compare their effect. As a measure of genotoxicity and cytotoxicity in cells, the micronucleus test will be used.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 and older
* good oral and general health
* non smokers

Exclusion Criteria:

* subjects suffering from infectious diseases or chronic inflammatory diseases
* use of antibiotics, corticosteroids and anti-inflammatory drugs in the last six months
* damage to the mucous membrane of the oral cavity
* subjects who have fixed-prosthetic works and orthodontic braces

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with cytotoxic and genotoxic effect of fluoridated toothpastes in buccal cells, assessed by micronucleus test | 90 days
  The micronucleus test is used to determine whether a compound is genotoxic by assessing the presence of micronuclei. Micronuclei can originate from chromosome fragments or whole chromosomes that cannot migrate to the poles during the anaphase phase of cell division. This test is widely used for monitoring buccal cells because of its precision for detecting chromosomal damage. The cells of the buccal mucosa will be taken with a cytological brush, the cell suspension is centrifuged, then applied to a microscope slide and fixed with methanol. The slides will be stained with Fast Green FCF dye and analyzed with an epifluorescence microscope.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No